CLINICAL TRIAL: NCT01439607
Title: Cellular and Molecular Mechanisms Governing Bone Marrow Stem Cells, Macrophages and Plasma Cell Biology in Gaucher Disease.
Brief Title: Cellular and Molecular Mechanisms Governing Bone Marrow Stem Cells in Gaucher Disease
Acronym: MGMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P081102
Record Dates: First submitted 2011-06-22; First posted 2011-09-23 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-04

CONDITIONS: Gaucher Disease
Keywords: Gaucher disease
MeSH Terms: conditions — Gaucher Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bone marrow and blood sampling (Experimental)
  Interventions: Other: Bone marrow and blood sampling

INTERVENTIONS:
Other: Bone marrow and blood sampling — Bone marrow and blood sampling

SUMMARY:
Gaucher disease is an inherited autosomal recessive lysosomal storage disorder caused by the defective activity of the glucocerebrosidase, leading to accumulation of glucocerebroside particularly in cells of the macrophage lineage. Clinical manifestations associate hematological, neurological and bone disorders.

DETAILED DESCRIPTION:
Gaucher disease is an inherited autosomal recessive lysosomal storage disorder caused by the defective activity of the glucocerebrosidase, leading to accumulation of glucocerebroside particularly in cells of the macrophage lineage. Clinical manifestations associate hematological, neurological and bone disorders.

In this project, the investigators aimed to study the cellular and molecular mechanisms governing the biology of various cell populations of the bone marrow and blood in these patients in order to define their potential role in the physiopathology of the disease. The main research topics the investigators plan will then be focused on characterization and functional analysis of hematopoietic stem cells, mesenchymal stem cells (with a special focus on osteogenic differentiation), macrophages and osteoclastic differentiation, B lymphocytes and plasma cells.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* Gaucher disease
* clinical examination written consent

Exclusion Criteria:

* pregnancy
* HIV seropositive
* contraindication to bone marrow sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-12; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
stem cells | day 1

CONTACTS AND LOCATIONS:
Overall Officials: Bertrabd Arnulf, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Bertrand Arnulf, Paris, Paris, France